CLINICAL TRIAL: NCT05963282
Title: Comparative Effectiveness of Entresto (Sacubitril/Valsartan) Versus ACEi/ARB in de Novo Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696B2037
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: de Novo Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Sacubitril/valsartan: Prescribed sacubitril/valsartan
- ACEi/ARB: Prescribed ACEi or ARB

SUMMARY:
This was a non-interventional retrospective cohort study of de novo heart failure with reduced ejection fraction (HFrEF) patients (aged ≥18 years) commencing first-line treatment on either sacubitril/valsartan or commencing or continuing angiotensin-converting enzyme inhibitors (ACEi)/angiotensin receptor blocker (ARB) therapy for HF in the United States (US) using the secondary source of data, Optum Electronic Health Records (EHR).

ELIGIBILITY:
Inclusion Criteria:

Sacubitril/valsartan cohort:

* Prescribed sacubitril/valsartan within the identification period.
* With at least one International Classification of Diseases, 9th Revision (ICD)-9 or 10th Revision (ICD-10) code for diagnosis of HF within 30 days prior to the index date (including index date), that had non-missing sex and year of birth data.
* Active in the database for 759 days prior to index.
* With left ventricular ejection fraction (LVEF) ≤ 40% known prior to index day (including index date).
* That were treated as part of the integrated delivery network (IDN).

ACEi/ARB cohort:

* Prescribed ACEi or ARB within the identification period.
* With at least one ICD-9 or ICD-10 code for diagnosis of HF within 30 days prior to the index date (including index date), that have non-missing sex and year of birth data.
* Active in the database for 759 days prior to index.
* With LVEF ≤ 40% known prior to index day (including index date).
* That were treated as part of the IDN.

Exclusion Criteria

Sacubitril/valsartan cohort:

* That were < 18 years old at index date.
* That were prescribed sacubitril/valsartan within the baseline period or identification period (whichever was earlier) at any time prior to the index date (excluding).
* With one or more ICD-9 or ICD-10 codes for diagnosis of HF within the baseline period, excluding the 30 days prior to index in which HF was initially identified (patient should have had no prior history of HF).
* That were prescribed ACEi/ARB > 2 days before index date, and within 30 days after a HF diagnosis during the identification period (i.e. any patient included in the ACEi/ARB cohort with an earlier index date, regardless of whether LVEF was ≤ 40% or > 40%)
* With LVEF ≤ 10% as the closest value to index date (including).

ACEi/ARB cohort:

* That were < 18 years old at index date.
* That were prescribed sacubitril/valsartan within the baseline period or identification period (whichever was earlier) at any time prior to the index date, on the index date, or until ≤ 2 days after the index date.
* With one or more ICD-9 or ICD-10 codes for diagnosis of HF within the baseline period, excluding the 30 days prior to index in which HF was initially identified (patient should have had no prior history of HF).
* With LVEF ≤ 10% as the closest value to index date (including).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 9870 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-19 (Actual)

PRIMARY OUTCOMES:
Total number of all-cause hospitalizations | Up to approximately 5 years

SECONDARY OUTCOMES:
Time to first all-cause hospitalization | Up to approximately 5 years
Number and proportion of HF-specific inpatient hospitalizations | Up to approximately 5 years
Number and proportion of HF-related inpatient hospitalizations | Up to approximately 5 years
Number and proportion of cardiovascular (CV)-specific inpatient hospitalizations | Up to approximately 5 years
Numbers and proportions of first and recurrent (1st, 2nd, 3rd, 4th and 5th) all-cause inpatient hospitalizations | Up to approximately 5 years
Numbers and proportions of first and recurrent (1st, 2nd, 3rd, 4th and 5th) HF-specific inpatient hospitalizations. | Up to approximately 5 years
Number and proportion of patients with ≥1 implantable cardioverter defibrillator (ICD) insertion during a hospitalization or during an emergency room (ER) visit for both the sacubitril/valsartan and ACEi/ARB cohorts | Up to approximately 5 years
Number and proportion of non-HF inpatient hospitalizations | Up to approximately 5 years
Number and proportion of non-CV inpatient hospitalizations | Up to approximately 5 years
Dosages and dose changes of sacubitril/valsartan administered | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States